CLINICAL TRIAL: NCT03670121
Title: A Pilot Study to Assess Treatment of Patients With Homogeneous Emphysema Using Sequential Segmental Bronchoscopic Thermal Vapor Ablation
Brief Title: A Pilot Study to Assess Treatment of Patients With Homogeneous Emphysema Using Sequential Segmental Bronchoscopic Thermal Vapor Ablation (NEXT STEP)
Acronym: NEXT STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uptake Medical Technology, Inc. (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-2346
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Emphysema or COPD
Keywords: COPD, Emphysema, Homogenous, Collateral Ventilation; Vapor; Ablation
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Single arm Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BTVA Treatment (Experimental): All patients that will receive Bronchoscopic Thermal Vapor Ablation (BTVA) Treatment
  Interventions: Device: Bronchoscopic Thermal Vapor Ablation (BTVA)

INTERVENTIONS:
Device: Bronchoscopic Thermal Vapor Ablation (BTVA) — Bronchoscopic vapor delivery to airway segment(s) targeted for treatment
  Other Names: BTVA; InterVapor

SUMMARY:
This study is a Prospective, single arm, single center pilot study following outcomes for 12 months after initial BTVA treatment. The primary objectives of the study are to prospectively document the safety and efficacy of sequential segmental treatment with BTVA in patients with a homogeneous distribution of emphysema that are not candidates for endobronchial valve therapy.

DETAILED DESCRIPTION:
The study will include patients with severe emphysema as defined by pulmonary function tests, a homogeneous distribution of emphysema as determined by CT, who are not eligible for endobronchial valve therapy based on fissure integrity as determined by CT. Enrollment will continue until 10 patients have been treated per protocol or until a maximum of 15 patients total have been treated.

Patients will be enrolled at Thoraxklinik University of Heidelberg, Germany and followed for twelve (12) months.

The follow up data collected will include pulmonary function testing (spirometry, body plethysmography, DLCO), exercise capacity (six minute walk test) and imaging findings (chest x-ray and CT). Dyspnea score (mMRC) and quality of life questionnaire (SGRQ-C) information will be obtained. Information regarding adverse events, serious adverse events, and major medical complications will be collected at each visit. Serious adverse events will be adjudicated by an independent medical monitor in order to establish relatedness to the InterVapor device and procedure.

Descriptive statistics will be used to summarize all safety and efficacy data. There is no predefined hypothesis regarding safety, or efficacy.

Monitoring of the study will be undertaken as a continuous process to ensure that high-quality data are obtained and to ensure compliance with study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or equal to 40 and ≤ 75 years old
2. At least one lung with a homogeneous distribution of emphysema (defined as a heterogeneity index < 1.2 when calculated as the ratio of upper lobe to lower lobe %-950 and when calculated as the ratio of lower lobe to upper lobe %-950) and a fissure integrity score < 95% as measured by CT
3. Contralateral lung (to lung targeted for the initial BTVA treatment) with tissue to air ratio > 8%
4. FEV1 between 20% and 45% predicted
5. TLC > or equal to 100% predicted
6. RV > or equal to 200% predicted
7. Post-rehabilitation 6MWD > 140 meters
8. Marked dyspnea scoring > or equal to 2 on the mMRC
9. Arterial blood gas levels of: PaCO2 ≤ 50 mm Hg; PaO2 > 45 mm Hg on room air
10. Non-smoking for 2 months prior to study enrollment, as confirmed by negative urine point of contact strips or serum cotinine level of ≤ 10 ng/mL, or negative CO Hb test
11. Optimized medical management (treatment consistent with GOLD guidelines)
12. Evidence of completed pulmonary rehabilitation:

    * ≥ 6 weeks out-patient or ≥ 3 weeks in-patient within 6 months of enrollment; or,
    * Patient has or continues to participate in regular physical activity beyond activities of daily living (i.e. a walking program) for ≥ 6 weeks with 6 months of enrollment under the supervision of a health care professional
13. Current influenza vaccination
14. Mentally and physically able to cooperate with the study procedures, follow-up requirements, and are able and willing to provide informed consent to participate in the study.

Exclusion Criteria:

1. Any condition that would interfere with the completion of the study, follow-up assessments, bronchoscopy, or that would adversely affect study outcomes. Concomitant illnesses or medications that would pose a significant increased risk for complications following treatment with BTVA. Relevant examples of relevance include immune system disorders, immunosuppressant medications of clinical relevance, bleeding disorders and unstable cardiovascular conditions, history of asthma or alpha-1 antitrypsin deficiency
2. DLCO < 20% predicted or immeasurable DLCO
3. BMI < 18kg/m2 or > 35 kg/m2
4. Clinically significant bronchiectasis with more than 30 ml productive cough
5. Heart and/or lung transplant, lung volume reduction surgery (LVRS), bullectomy, or thoracic surgery with removal of lung tissue
6. Prior lung volume reduction via endobronchial valves(s), stent(s), coil(s), and/or polymer. Patients whose endobronchial valves have been removed can be treated if: all valves removed ≥ 6 months prior to BTVA and baseline bronchoscopy reveals no airway obstruction or obvious tissue granulation
7. Recent respiratory infections or COPD exacerbation in preceding 6 weeks
8. Unstable COPD (any of the following):

   * >3 COPD related hospitalizations requiring antibiotics in past 12 months
   * COPD related hospitalization in past 3 months
   * daily use of systemic steroids, i.e. > 5 mg prednisolone
9. Single large bulla (defined as > 1/3 volume of the lobe) or a paraseptal distribution of emphysema in lobe to be treated
10. Bacterial infection or symptoms indicative of active infection (i.e., fever, elevated white blood cell count)
11. History of any of the following:

    * Left ventricular ejection fraction (EF) ≤ 40%
    * Stroke
    * Myocardial infarction or acute coronary syndrome in previous year
    * Current use of anticoagulants (including warfarin, and NOACs such as dabigatran, rivaroxaban, apixaban, and similar).
    * Patient is unable to stop antiplatelet therapy (including dipyridamole, clopidogrel, prasugrel, and ticlopidine) 7 days before and not restart until 7 days after study procedure.
    * Known sensitivity to medications required to perform bronchoscopy
12. Pulmonary hypertension:

    * Peak systolic PAP > 45 mm Hg or
    * Mean PAP > 35 mm Hg
    * Right heart catheter measurements (if available) will be considered definitive over echocardiography or cardiac scintigraphy measurements
13. Newly prescribed morphine derivatives within the last 4 weeks
14. Pregnant or breastfeeding
15. Pneumothorax or pleural effusion within previous 6 months
16. Indwelling pacemaker or implantable cardiac defibrillator (ICD)
17. Patients dependent on the sponsor or investigator
18. Current enrollment in any other investigational study which has not completed requisite follow-up

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence of SAEs, Major Medical complications, and unanticipated serious adverse device effects (USADEs) (safety endpoint) | Baseline to 6 months
  Occurrence of SAEs, Major Medical complications, and unanticipated serious adverse device effects (USADEs) (safety endpoint)
Change in FEV1 (efficacy endpoint) | Baseline to 6 months
  Change in FEV1 (efficacy endpoint)
Change in St Georges Respiratory Questionnaire for COPD Patients (SGRQ-C) score (efficacy endpoint) | Baseline to 6 months
  This trial will utilize the SGRQ-C which is a shortened version of the SGRQ questionnaire. The SGRQ is a validated, disease-specific questionnaire that measures health-related quality of life in patients with COPD.
  The instrument has 3 domains (activity, symptoms, and impacts) and a total score. A Total and three-component scores are calculated: Symptoms; Activity; Impacts. Each questionnaire response has a unique empirically derived 'weight'. The lowest possible weight is zero and the highest is 100. Each component of the questionnaire is scored separately. Sum of maximum possible weights for each component and Total: Symptoms 566.2, Activity 982.9, Impacts 1652.8. Total (sum of maximum for all three components) 3201.9 Higher weights indicate worse outcomes. The difference in the domain scores and total score at follow-up visits relative to baseline will be calculated and reported.

SECONDARY OUTCOMES:
Change in FVC | Baseline to 6 months
  Change in Forced Vital Capacity
Change in FRC | Baseline to 6 months
  Change in Forced Residual Capacity
Change in RV | Baseline to 6 months
  Change in Residual Volume
Change in TLC | Baseline to 6 months
  Change in Total Lung Capacity
Change in RV/TLC | Baseline to 6 months
  Change in Residual Volume/Total Lung Capacity
Change in DLCO | Baseline to 6 months
  Change in Diffusing capacity of the lung for carbon monoxide
Change in Modified Medical Research Council (mMRC) Dyspnea scale | Baseline to 6 months
  Change in dyspnea score.
  Grade Degree of Breathlessness Related to Activities Grade 0 No breathlessness except with strenuous exercise Grade 1 Breathlessness when hurrying on the level or walking up a slight hill Grade 2 Walks slower than people of the same age on the level because of breathlessness or has to stop for breath when walking at own pace on the level Grade 3 Stops for breath after walking about 100 yards or a few minutes on the level Grade 4 Too breathless to leave the house or breathless when dressing or undressing Max score=4, Min score=0 One score is reported based on grade. Higher values represent worse outcomes. For patients with a higher mMRC grade (e.g. ≥2) and clinical circumstances consistent with respiratory disease, measuring spirometry (e.g., FEV₁ and FVC), determining the patient's GOLD stage, helps guide therapeutic interventions.
Change in 6MWD | Baseline to 6 months
  Change in six minute walk distance
Change in volume of the treated lobe(s) | Baseline to 6 months
  Change in lung volume assessed by CT

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, Principal Investigator — Univ.-Prof. Felix JF Herth, Thoraxklinik University of Heidelberg Heidelberg, Germany
Locations (1):
- Thoraxklinik University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989